Title: ABCA3 gene and RDS in late preterm and term infants

NCT number: NCT04137783

**Date of document:** March 16, 2021

Neonatal respiratory distress syndrome (RDS) is caused by the deficiency or inactivation of pulmonary surfactant, and is commonly seen in early preterm infants due to their immature lung development. However, some maternal and neonatal characteristics in late preterm and term infants such as maternal diabetes, meconium aspirated pneumonia, neonatal sepsis, and severe intrapartum asphyxia, could also contribute to RDS. Existing evidence has demonstrated that RDS in late preterm and term infants is a somewhat distinct disease entity, with risk factors and clinical profiles that differ from those in early preterm infants [1-3]. In a neonatal unit, some late preterm or term infants experience RDS; however, the etiology has not been well defined after a routine workup. This unique RDS entity was referred to as unexplained respiratory distress syndrome (URDS) by numerous previous studies, as well as our study [4-7].

Given that a large body of literature has demonstrated the essential role genetic mechanism play in the pathogenesis of most URDS cases, numerous medical facilities have carried out clinical exome sequencing to identify the underlying genetic cause of URDS [8-10]. Among all of the genetic factors that contribute to the RDS, the most common is *ABCA3* gene mutation, which involves the assembly of pulmonary surfactant in the lamellar body of pneumocyte II [11]. Existing evidence indicated that patients with homozygous or compound heterozygous *ABCA3* gene mutations were commonly in critically ill conditions [12]. A single *ABCA3* mutation was also likely to increase the risk and severity of RDS [4, 13].

Unfortunately, in a considerable proportion of neonatal URDS patients, genetic testing fails to yield any abnormal findings, making these patients the "true URDS" patients. Currently, whether the *ABCA3*-mutated URDS patients have similar or more challenging clinical profiles to those without any genetic abnormalities continues to confound most neonatologists. An answer to this question would help to guide the management and predict

the clinical outcomes of neonatal URDS patients. The present study aimed to address this by comparing the clinical characteristics of late preterm and term infants with severe URDS with homozygous or compound heterozygous *ABCA3* mutations, a single *ABCA3* mutation, or no defined genetic abnormalities.

#### **Patient selection**

This single-center retrospective cohort study involved infants  $\geq$  34 weeks' gestation with severe URDS who were admitted to Children's Hospital of Chongqing Medical University between January 2013 and December 2019. In this study, severe RDS was mainly defined according to the consensus of the Pediatric Acute Lung Injury Consensus Conference [14], and Montreux definition [15]: (1) manifestations and chest radiograph compatible with RDS; (2) on invasive mechanical ventilation with oxygenation index  $\geq$  16, which was calculated based on the daily blood gas, or as an alternative measurement, on the subcutaneous oxygen tension [16,17]

Almost all infants with severe RDS had undergone a comprehensive workup, including serial infection markers, chest radiograph, echocardiography, and blood and sputum pathogen testing. For all patients with severe RDS who responded inadequately to interventions and had unremarkable workup findings, trio exome sequencing on samples from patients and their parents were usually recommended. All URDS patients who underwent genetic testing were enrolled in this study. Those whose parents rejected genetic testing, or who had cardiopulmonary malformations, pulmonary hypoplasia, culture-positive sepsis, or known respiratory disease-associated gene mutations (such as SFTPA1, SFTPA2, SFTPB, SFTPC, CHPT1, LPCAT1, PCYT1B, NKX2, CFTR, and FOXF1) were excluded. This study was approved by the Institutional Review Board of Children's Hospital of the Chongqing Medical University (No.2018-158) and was registered on clinicaltrials.gov (NCT04137783).

#### **Exome sequencing and gene mutation detection**

All infants in this study underwent trio exome sequencing after written consent had been obtained from their parents. A gene company (Chigene, Beijing) offered the sequencing as a clinical laboratory service. Sequence analysis of coding exons and flanking introns were performed as previously described [18,19]. All samples were analyzed to detect frame-shift mutations, nonsense mutations, missense mutations, splicing site mutations, and in-frame indel mutations. Assessment of copy number variation was also performed from exome sequencing data using computational tools. A variant was strictly defined as a mutation if it had been previously described to cause disease with a presentation consistent with these patients, or resulted in an amino acid change or protein structure alteration to disrupt protein function that was predicted by both SIFT and PolyPhen for missense mutations [20, 21], and MaxEntScan and dbscSNV for splicing site mutations<sup>[22]</sup>. In the case of a novel mutation, phastCons and phyloP were used to determine the evolutionary conservation of the region where the mutation was located [23]. The American College of Medical Genetics and Genomics/Association for Molecular Pathology (ACMG-AMP) criteria were applied to interpret the mutations [24]. The subjects in this study were categorized into three groups: homozygous or compound heterozygous ABCA3 mutations, a single ABCA3 mutation, and no defined genetic abnormalities.

## Clinical profiles data

All relevant clinical data were extracted from a hospital information system.

All antepartum and postpartum data were collected and included: maternal age, parity, and pregnancy-related complications; mode of birth, amniotic fluid condition, and history of asphyxia and resuscitation; postnatal age of respiratory symptom onset, modalities of respiratory support, and the daily record of blood gas and subcutaneous oxygen tension; laboratory data including complete blood count, C-reactive protein, procalcitonin, blood and sputum culture, respiratory viral detection test, and genetic testing; radiographic examination including chest X-ray and echocardiogram; medications taken during the hospital stay.

### Radiological scoring

All chest X-rays were reviewed on a hospital information system by one radiologist. The most severe images were scored according to the Fleischner Society criteria<sup>[25]</sup>. The chest X-ray was rated in three sections on both sides of the lung: apex to the carina, carina to the lower pulmonary vein, and lower pulmonary vein to the diaphragm. The incidence of radiological features, including ground-glass opacity, reticular pattern, air bronchogram, atelectasis, and air leak, were evaluated for each lung section. Each finding was scored as 0 = none, 1 = discrete, 2 = diffuse, or 3 = strong at each section. An overall cumulative score was calculated by adding the individual section scores together, with a maximum score of 18 for each patient.

# **Statistical Analysis**

Analysis of variance (ANOVA) and the Chi-square or Fisher's exact tests were used to compare clinical characteristics and radiographic scores between different groups of patients. Tests for the differences in the age of symptom onset and the age of development of severe RDS between the groups were carried out using the log-rank test. A two-tailed *p*-value of

#### References

- [1]. Wang J, Liu X, Zhu T, et al. Analysis of neonatal respiratory distress syndrome among different gestational segments. Int J Clin Exp Med 2015; 8:16273-9.
- [2]. Shi Y, Tang S, Zhao J, et al. A prospective, randomized, controlled study of NIPPV versus nCPAP in preterm and term infants with respiratory distress syndrome. Pediatr Pulmonol 2014; 49:673-8.
- [3].Condò V, Cipriani S, Colnaghi M, et al. Neonatal respiratory distress syndrome: are risk factors the same in preterm and term infants?. J Matern Fetal Neonatal Med 2017; 30:1267-72.
- [4]. Somaschini M, Presi S, Ferrari M, et al. Surfactant proteins gene variants in premature newborn infants with severe respiratory distress syndrome. J Perinatol 2018; 38:337-44.
- [5].Brasch F, Schimanski S, Mühlfeld C, et al. Alteration of the pulmonary surfactant system in full-term infants with hereditary ABCA3 deficiency. Am J Respir Crit Care Med 2006; 174:571-80.
- [6].Guala A, Carrera P, Pastore G, et al. Familial clustering of unexplained transient respiratory distress in 12 newborns from three unrelated families suggests an autosomal-recessive inheritance. Scientific World Journal 2007; 7:1611-6.
- [7]. Somaschini M, Nogee LM, Sassi I, et al. Unexplained neonatal respiratory distress due to congenital surfactant deficiency. J Pediatr 2007; 150:649-53.
- [8]. Shen CL, Zhang Q, Meyer J, et al. Genetic Factors Contribute to Risk for Neonatal Respiratory Distress Syndrome among Moderately Preterm, Late Preterm, and Term Infants. J Pediatr 2016; 172:69-74.e2.
- [9]. Schindlbeck U, Wittmann T, Hoppner S, et al. ABCA3 missense mutations causing surfactant dysfunction disorders have distinct cellular phenotypes. Hum Mutat 2018; 39:841-50.
- [10].Bhandari V. Bronchopulmonary dysplasia. New Jersey: Springer; 2016
- [11].Besnard V, Matsuzaki Y, Clark J, et al. Conditional deletion of ABCA3 in alveolar type II cells alters surfactant homeostasis in newborn and adult mice. Am J Physiol Lung Cell Mol Physiol 2010; 298:L646-59.
- [12]. Wambach JA, Casey AM, Fishman MP, et al. Genotype-phenotype correlations for infants and children with ABCA3 deficiency. Am J Respir Crit Care Med 2014; 189:1538-43.
- [13]. Wambach JA, Wegner DJ, Depass K, et al. Single ABCA3 mutations increase risk for neonatal respiratory distress syndrome. Pediatrics 2012; 130:e1575-82.
- [14].Khemani RG, Smith LS, Zimmerman JJ, et al. Pediatric acute respiratory distress syndrome: definition, incidence, and epidemiology: proceedings from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med 2015; 16:S23-S40.
- [15].De Luca D, van Kaam AH, Tingay DG, et al. The Montreux definition of neonatal ARDS: biological and clinical background behind the description of a new entity. Lancet Respir Med 2017; 5:657-66.
- [16].Rooth G, Huch A, Huch R. Transcutaneous oxygen monitors are reliable indicators of arterial oxygen tension (if used correctly). Pediatrics 1987; 79:283-6.
- [17].Sandberg KL, Brynjarsson H, Hjalmarson O. Transcutaneous blood gas monitoring during neonatal intensive care. Acta Paediatr 2011; 100:676-9.
- [18].Li L, Deheragoda M, Lu Y, et al. Hypothyroidism Associated with ATP8B1 Deficiency. J Pediatr 2015; 167:1334-9.e1.
- [19].Meng L, Pammi M, Saronwala A, et al. Use of Exome Sequencing for Infants in Intensive Care Units: Ascertainment of Severe Single-Gene Disorders and Effect on Medical Management. JAMA Pediatr 2017; 171:e173438.
- [20].Kumar P, Henikoff S, Ng PC. Predicting the effects of coding non-synonymous variants on protein function using the SIFT algorithm. Nat Protoc 2009; 4:1073-81.
- [21]. Adzhubei IA, Schmidt S, Peshkin L, et al. A method and server for predicting damaging missense mutations. Nat Methods 2010; 7:248-9.
- [22].Sexton CE, Wadsworth ME, Miller JB, et al. Splice Site Variant Analyzer: Determining the Pathogenicity of Splice Site Variants. J Biomed Res Prac 2018; 2:100012.
- [23].Ramani R, Krumholz K, Huang YF, et al. PhastWeb: a web interface for evolutionary conservation scoring of multiple sequence alignments using phastCons and phyloP.

- Bioinformatics 2019; 35:2320-2.
- [24].Richards S, Aziz N, Bale S, et al. Standards and guidelines for the interpretation of sequence variants: a joint consensus recommendation of the American College of Medical Genetics and Genomics and the Association for Molecular Pathology. Genet Med 2015;17:405-23.
- [25].Hansell DM, Bankier AA, Macmahon H, et al. Fleischner Society: glossary of terms for thoracic imaging. Radiology 2008; 246:697-722.